CLINICAL TRIAL: NCT04835532
Title: Tenting Screws in Combination With Platelet Concentrate for Vertical Alveolar Ridge Augmentation: Prospective, Blinded, Randomized Controlled Trial
Brief Title: Tenting Screws in Combination With Platelet Concentrate for Vertical Alveolar Ridge Augmentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-0050
Record Dates: First submitted 2021-03-16; First posted 2021-04-08 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-02

CONDITIONS: Bone Loss, Alveolar
Keywords: tenting screws; advanced platelet rich fibrin; injectable platelet rich fibrin; guided bone regeneration
MeSH Terms: conditions — Alveolar Bone Loss | interventions — proliferation regulatory factors, human urine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Experimental): Vertical alveolar bone augmentation was performed by GBR technique before implantation.
  BIO-OSS+ BIO-GIDE barrier membrane
  Interventions: Procedure: guided bone gereration
- Treatment group 1 (Experimental): Vertical alveolar bone augmentation was performed by GBR technique and tenting screws before implantation.
  BIO-OSS+ BIO-GIDE barrier membrane+ tenting screws
  Interventions: Procedure: guided bone gereration
- Treatment group 2 (Experimental): Vertical alveolar bone augmentation was performed by GBR technique in combination with tenting screws and A-PRF, I-PRF before implantation.
  BIO-OSS+ BIO-GIDE barrier membrane+ tenting screws+A-PRF, I-PRF
  Interventions: Procedure: guided bone gereration

INTERVENTIONS:
Procedure: guided bone gereration — guided bone generation: GBR is a procedure that uses barrier membranes with or without particulate bone grafts or/and bone substitutes.
  tenting screws: Screws are implanted in the surgical area to prevent the barrier membrane from collapsing.
  A-PRF/I-PRF: Obtained by autologous blood centrifugation.
  Other Names: tenting screws, A-PRF, I-PRF

SUMMARY:
Alveolar bone resorption often occurs after tooth extraction. At present, guided bone regeneration technique is widely used in clinic since it leads to less trauma and less complications. Tenting screw technology, basic on the classical GBR, implants screws into the surgical area to prevent the barrier membrane from collapsing. Moreover, advanced platelet rich fibrin and injectable platelet-rich fibrin are used to provide the osteogenic function. The investigators intend to increase vertical alveolar bone augmentation by combining tenting screws and A-PRF, I-PRF.

DETAILED DESCRIPTION:
Alveolar bone resorption often occurs after tooth extraction. At present, guided bone regeneration technique is widely used in clinic since it leads to less trauma and less complications. Tenting screw technology, basic on the classical GBR, implants screws into the surgical area to prevent the barrier membrane from collapsing. Moreover, advanced platelet rich fibrin and injectable platelet-rich fibrin are used to provide the osteogenic function. The investigators intend to increase vertical alveolar bone augmentation by combining tenting screws and A-PRF, I-PRF.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old;
2. single tooth in the maxillary posterior area cannot be retained (third degree loosening / alveolar bone resorption to the periapical area), implantation is needed after extraction, and CBCT shows vertical bone defect ≥ 3mm;
3. 4 weeks after extraction or missing teeth within 3-5 weeks;
4. adjacent teeth exist and loosening is less than Ⅰ degree;
5. periodontal disease in inactive stage, whole mouth bleeding index (FMBS) is less than 20%;
6. thick gingival biological type.
7. CBCT shows that the bone of the edentulous site meets the requirements of tent screw implantation (bone height ≥ 3mm and bone mineral density is sufficient);
8. the patients and their families have informed consent and signed the informed consent form.

Exclusion Criteria:

1. pregnant and lactating women;
2. smoking (> 10 cigarettes per day) and alcoholism;
3. taking anticoagulants within 3 months before operation;
4. suffering from autoimmune diseases, diabetes, liver disease, blood system diseases and infectious diseases;
5. patients taking any drugs that affect platelet function or whose platelet count is less than 200000/mm3 3 months before blood collection;
6. patients who have been treated with bisphosphate / steroids for a long time;
7. have received alveolar ridge bone augmentation surgery;
8. previous history of radiotherapy in the head and neck;
9. acute inflammation in edentulous sites;
10. inability to maintain good oral hygiene or follow-up visits as required.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Buccal bone augmentation, BBA(bone height changes between T0 and T2) | T0(before surgery), T2(6 months after GBR)
  The sagittal plane of CBCT image is selected as the measuring plane, and the horizontal tangent of the inferior margin of maxillary sinus / paranasal sinus is selected as the baseline. The investigaters will measure the bone height changes by CBCT(three-dimensional CT) and Related measurement software. The unit of measurement is millimeter.

SECONDARY OUTCOMES:
Lingual bone augmentation, LBA(bone height changes between T0 and T2) | T0(before surgery), T2(6 months after GBR)
  The sagittal plane of CBCT image is selected as the measuring plane, and the horizontal tangent of the inferior margin of maxillary sinus / paranasal sinus is selected as the baseline.
  The sagittal plane of CBCT image is selected as the measuring plane, and the horizontal tangent of the inferior margin of maxillary sinus / paranasal sinus is selected as the baseline.The investigaters will measure the bone height changes by CBCT(three-dimensional CT) and Related measurement software. The unit of measurement is millimeter.

OTHER OUTCOMES:
Bone density, BD | T2(6 months after GBR)
  in the area of bone regeneration, ranging 2mm × 2mm

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No